CLINICAL TRIAL: NCT05063110
Title: Treatment of Non Severe Hemophagocytosis Lymphohistiocytosis With ITACITINIB a Phase II Prospective Trial
Brief Title: Treatment of Non Severe Hemophagocytosis Lymphohistiocytosis With ITACITINIB
Acronym: HLH-JAK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP 201454; 2021-000407-20 (EudraCT Number)
Record Dates: First submitted 2021-09-02; First posted 2021-09-30 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-10

CONDITIONS: Adults Patients Having Non Severe HLH
Keywords: Hemophagocytosis lymphohistiocytosis; JAK 1; Itacitinib
MeSH Terms: interventions — itacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): 300 mg of ITACITINIB will be administrated per os every day for 30 days, dose with reduction to 200 mg per safety is allowed if AEs are observed or if co-administered a strong CYP3A inhibitor
  Interventions: Drug: Itacitinib

INTERVENTIONS:
Drug: Itacitinib — Administration of 300 mg of ITACITINIB per os every day for 30 days.

SUMMARY:
This project aims to test the effectiveness of ITACITINIB in sporadic Hemophagocytosis Lymphohistiocytosis (HLHs)

DETAILED DESCRIPTION:
This project aims to test the effectiveness of ITACITINIB in sporadic Hemophagocytosis Lymphohistiocytosis (HLHs). The existence of an IFN-γ signature, in HLHs, is a strong rational for testing the use of a JAK1 inhibitor in the treatment of HLHs. We hypothesize that ITACITINIB, an inhibitor of JAK-1, may be a therapeutic of interest in the treatment of non-severe HLHs in replacement of corticosteroids by inhibiting the production and effects of IFN-γ but also those of other pro-inflammatory cytokines. The use JAK-1 inhibitor instead of corticosteroids in patients with HLHs without any sign of severity is justified by its probable lesser toxicity and higher efficiency.

In this proof of concept study, because of the vital risk associated with severe HLH and the efficacy of Etoposide in this setting, we will first include only patients with moderate HLHs

ELIGIBILITY:
Inclusion Criteria:

* Patients age > 18 years,
* Patient is willing to provide written informed consent prior to enrolment and agrees to follow the protocol
* Patient known to have systemic juvenile idiopathic arthritis are classified as having HLH
* Negative pregnancy test for woman of childbearing potential, woman of childbearing potential should have reliable contraception for the duration of the study
* Be either affiliated to, or a beneficiary of, a social security category

Exclusion Criteria:

* Organ failure: confusion, organic kidney failure KDIGO 2 criteria, liver failure (Factor V < 50%), heart failure, respiratory failure.
* Fibrinogen < 0.50 g/l, platelets <20G/L
* Indication to intensive care unit transfer on an organ failure requiring assistance (dialysis, Ventilation (assisted or VNI), shock regardless of the origin.
* Breastfeeding women
* Patient participating in another investigational therapeutic study
* Women with a positive pregnancy test or not willing to take contraceptive measures
* Known allergies, hypersensitivity, or intolerance to any of the ITACITINIB or excipients, or similar compounds
* Current or history of recurrent infections, including HBV, HCV
* Participants with active HBV or HCV infection that requires treatment or who are at risk for HBV reactivation (ie Positive HBs Ag serology)
* Candidates positive for HCV antibody and positive PCR RNA HCV
* HIV infection with positive viral charge
* Protected adults (including individual under guardianship by court order)
* Vulnerable adults, under a safeguard of justice measure
* Adults deprived of their liberty by judicial or administrative decision
* Persons under psychiatric care without their consent
* Persons admitted to social institution for purposes other this research
* Adults under legal protection (guardianship or curatorship)
* Persons unable to express their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of ITACITINIB | At day 15
  Efficacy at day 15 of ITACITINIB treatment in non-severe adults HLH

SECONDARY OUTCOMES:
Response rate of ITACITINIB at D8 on clinical and biological symptoms of primitive/refractory/relapse adults HLHs without severity criteria | day 8
  Response rate at D8 of treatment
Efficacy at the day of etiologic treatment if patients received at least 7 days of treatment (ITACITINIB taken until J15) | At day 15
  Rate of complete response to ITACITINIB treatment for HLHs in adults without any sign of severity at the day of etiologic treatment if patients have been treated by ITACITINIB at least during seven days. Response to ITACITINIB is evaluated at the day of etiologic treatment on the major and minor diagnostic criteria of HLH
Toxicity of ITACITINIB | 21 months
  Toxicity of ITACITINIB not related to evolution of HLH (cytopenia, worsening of hepatic balance, secondary infections)
Rescue therapy | 21 months
  In the case of worsening, treatment will be stopped and switch for HLH specific treatment as VP16, (etoposide)
Reduction of plasma cytokines level between D0 and D15 and correlation to the therapeutic response to D15 | At day 15
  Range of decrease in plasma rate of IFN-Gamma, IP-10, Il-1, Il-6, IL-10, TNF-alpha, between D0 and D15 of ITACITINIB treatment in each patient group: response and progression
Clinical, biological, associated diseases characteristics of patients having CR, PR, Progression | 21 months
  Clinical, biological, associated diseases and evolutions characteristics of patients in each response
Overall survival at 3 | 3 months
  Overall survival at 3
Response rate of ITACITINIB at D30 on clinical and biological symptoms of primitive/refractory/relapse adults HLHs without severity criteria | day 30
  Response rate at D30 of treatment
Response rate of ITACITINIB at D90 on clinical and biological symptoms of primitive/refractory/relapse adults HLHs without severity criteria | day 90
  Response rate at D90 of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Avicenne, Bobigny, Bobigny, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Menasche G, Feldmann J, Fischer A, de Saint Basile G. Primary hemophagocytic syndromes point to a direct link between lymphocyte cytotoxicity and homeostasis. Immunol Rev. 2005 Feb;203:165-79. doi: 10.1111/j.0105-2896.2005.00224.x. PMID 15661029
- [Result] Pachlopnik Schmid J, Ho CH, Chretien F, Lefebvre JM, Pivert G, Kosco-Vilbois M, Ferlin W, Geissmann F, Fischer A, de Saint Basile G. Neutralization of IFNgamma defeats haemophagocytosis in LCMV-infected perforin- and Rab27a-deficient mice. EMBO Mol Med. 2009 May;1(2):112-24. doi: 10.1002/emmm.200900009. PMID 20049711
- [Result] Billiau AD, Roskams T, Van Damme-Lombaerts R, Matthys P, Wouters C. Macrophage activation syndrome: characteristic findings on liver biopsy illustrating the key role of activated, IFN-gamma-producing lymphocytes and IL-6- and TNF-alpha-producing macrophages. Blood. 2005 Feb 15;105(4):1648-51. doi: 10.1182/blood-2004-08-2997. Epub 2004 Oct 5. PMID 15466922
- [Result] Vainchenker W, Constantinescu SN. JAK/STAT signaling in hematological malignancies. Oncogene. 2013 May 23;32(21):2601-13. doi: 10.1038/onc.2012.347. Epub 2012 Aug 6. PMID 22869151
- [Result] Maschalidi S, Sepulveda FE, Garrigue A, Fischer A, de Saint Basile G. Therapeutic effect of JAK1/2 blockade on the manifestations of hemophagocytic lymphohistiocytosis in mice. Blood. 2016 Jul 7;128(1):60-71. doi: 10.1182/blood-2016-02-700013. Epub 2016 May 24. PMID 27222478